CLINICAL TRIAL: NCT01652794
Title: A Phase 1 Study of Carboplatin and Gemcitabine Chemotherapy and Stereotactic Body Radiosurgery for the Palliative Treatment of Persistent or Recurrent Gynecologic Cancer
Brief Title: Carboplatin, Gemcitabine Hydrochloride, and Stereotactic Body Radiation Therapy in Gynecological Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE8810; NCI-2012-00608 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Leydig Cell Tumor; Ovarian Sarcoma; Ovarian Stromal Cancer; Pseudomyxoma Peritonei; Recurrent Cervical Cancer; Recurrent Endometrial Carcinoma; Recurrent Fallopian Tube Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Primary Peritoneal Cavity Cancer; Recurrent Uterine Sarcoma; Recurrent Vaginal Cancer; Recurrent Vulvar Cancer
MeSH Terms: conditions — Leydig Cell Tumor; Pseudomyxoma Peritonei; Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Radiosurgery; Carboplatin; Gemcitabine; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (carboplatin, gemcitabine hydrochloride, and SBRT) (Experimental): Patients also receive carboplatin IV over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on day 1 and undergo SBRT on days 2-4.
  Interventions: Radiation: stereotactic body radiation therapy; Drug: carboplatin; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis; Other: pharmacogenomic studies

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — Undergo SBRT
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: laboratory biomarker analysis — Optional correlative studies
Other: pharmacogenomic studies — Optional correlative studies
  Other Names: Pharmacogenomic Study

SUMMARY:
The purpose of this phase I study is to determine the highest dose of carboplatin and gemcitabine (gemcitabine hydrochloride) that can be given safely to subjects with gynecologic cancer, in combination with stereotactic body radiation therapy (SBRT). This dose is called the maximum tolerated dose (MTD). To determine the MTD, patients will receive different amounts of carboplatin and gemcitabine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine maximum tolerated carboplatin/gemcitabine dose administered with SBRT as measured by < 30-day acute toxicity defined by Common Terminology Criteria for Adverse Events (CTCAE) v4.0.

SECONDARY OBJECTIVES:

I. Off-study SBRT target local control assessment: 6-week post-trial fludeoxyglucose F 18 (18F-FDG) positron emission tomography (PET)/computed tomography (CT) or other imaging response by European Organisation for Research and Treatment of Cancer (EORTC) PET criteria as listed and National Cancer Institute (NCI) guidelines.

II. Off-treatment late toxicity assessment: record 3-month and 6-month radiation-related toxicity defined by CTCAE v4.0.

III. Off-study global clinical benefit assessment: 6-month post-therapy clinical benefit (defined as percentage of patients who had complete, partial, or stable disease for at least 6 months).

TERTIARY OBJECTIVES:

I. Associate pretherapy tumor biopsy ribonucleotide reductase (R1, R2, p53R2), Tip60 and Poly(ADP-ribose) polymerase 1/2 expression with 6-week therapy response.

OUTLINE: This is a dose-escalation study of carboplatin and gemcitabine hydrochloride.

Patients also receive carboplatin intravenously (IV) over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on day 1 and undergo SBRT on days 2-4.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 1 year, and then yearly for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient has diagnosis of a persistent or recurrent gynecologic cancer
* Patient age is > 18 years.
* Patient must have at least one abdominopelvic measurable site of disease as defined by 9.1.3;. A treatment planning 18F-FDG positron emission tomography and computed tomography scan (PET/CT; whole body) may be used to complement assessment, & if done must be completed prior to first dose of carboplatin / gemcitabine and within 35 days of first day of SBRT. There MUST BE no more than four (4) intended radiosurgical target lesions. An individual (one of up to four) radiosurgical target lesion MUST NOT EXCEED a volume of no greater than 160 cubic centimeters (cc).
* No prior cryosurgery or radiofrequency ablation in SBRT-target lesion. Patients with prior cryoablation and radiofrequency ablation are excluded as these treatments are designed to destroy tissue with freezing or heat. Radiation treatments given by SBRT may not work biologically or may cause excessive tissue injury in patients who have had prior cryoablation and radiofrequency ablation.
* Patient has no major medical illnesses or psychiatric illnesses:

  1. New York Heart Association (NYHA) class 3 or 4 congestive heart failure;
  2. unstable angina pectoris;
  3. symptomatic cardiac arrhythmia;
  4. hypertension with diastolic blood pressure greater than 110 mmHg;
  5. pulmonary disease consisting of dyspnea at rest requiring oxygen supplementation;
  6. renal function impairment (defined here as baseline serum creatinine >2.0 mg/dL);
  7. psychiatric illness/social situations that would limit compliance.
* Patient must have no known brain metastases. These patients are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound neurological and other adverse event evaluation.
* Patient must demonstrate adequate organ function (< 35 days from enrollment):

  * Bone marrow: absolute neutrophil count (ANC) ≥ 1500/mcl, platelets ≥ 100,000, hemoglobin ≥ 10 mg/dL.
  * Renal function: creatinine ≤ 2.0 mg/dL.
  * Hepatic function: bilirubin ≤ 1.5X institutional upper limit of normal (ULN); AST, ALT, alkaline phosphatase ≤ 2.5X ULN
* Patient MUST have had prior chemotherapy or radiation for a gynecologic cancer. Patient is > 28 days from previous treatment (chemotherapy or radiation) and toxicities related to the previous treatment must have resolved to grade 1 or baseline.
* Patient has Gynecologic Oncology Group performance status score of 0 or 1.
* Patient is able to give study-specific informed consent

Exclusion Criteria:

* Any patient NOT meeting the above criteria
* Any patient with active connective tissue disease such as lupus or dermatomyositis is excluded; patients with active connective tissue disease are at an excessive risk of organ function-impairing fibrosis
* Any patient with active Crohn's disease or active ulcerative colitis is excluded; patients having these conditions are at an excessive risk of organ function-impairing fibrosis
* Any patient with known anaphylaxis to carboplatin or gemcitabine is excluded
* Pregnant women are excluded from this study because radiation has the potential for teratogenic or abortifacient effects; screening beta-human chorionic gonadotropin (hcg) levels (urine or blood) and diagnostic tests will be used to determine eligibility in women of childbearing potential; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; these potential risks may also apply to carboplatin/gemcitabine chemotherapy agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with carboplatin or gemcitabine; in addition, patients known to be HIV-positive patient are excluded due to an increased risk of lethal infections when treated with marrow-suppressive therapy such as carboplatin/gemcitabine; HIV testing is not mandatory for eligibility evaluation
* Due to a perceived increased risk to transplanted organ for lethal dysfunction or lethal infection, patients with visceral organ transplants are not eligible
* Patients with other active non-gynecologic invasive malignancies are excluded; patients with other invasive malignancies who had (or have) cancer present within the last two years are excluded

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Rate of acute grade 3-5 toxicities following carboplatin/gemcitabine hydrochloride and SBRT treatment graded based on CTCAE, version 4.0 | Within 30 days of completing treatment
  A modified Fibonacci design used during the dose-finding portion of this study. When =< 1 out of 6 patients enter at highest next dose level below the maximum tolerated dose (MTD), this is the recommended phase 2 dose. At least 6 patients must be entered at the recommended phase 2 dose.

SECONDARY OUTCOMES:
Progression-free survival | From the time from registration until time of progression, recurrence, or death, up to 6 months
  Calculated following the method of Kaplan and Meier and survival dependence on measured covariates will be assessed using the Cox proportional hazards model.
Survival dependence on measured covariates | Up to 5 years
  Descriptive and tabular data will be reported. Assessed using the Cox proportional hazards model.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Waggoner, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States